CLINICAL TRIAL: NCT01090713
Title: Lisdexamfetamine in Binge Eating Disorder of Moderate or Greater Severity
Brief Title: Efficacy Study of Lisdexamfetamine to Treat Binge Eating Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Collaborators: Shire (Industry); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LDX in BED
Record Dates: First submitted 2010-03-19; First posted 2010-03-22 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lisdexamfetamine (Active Comparator): drug
  Interventions: Drug: lisdexamfetamine
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: lisdexamfetamine — oral; 20-70mg/day
  Arms: Lisdexamfetamine
Drug: Placebo control — 20-70mg; oral
  Arms: Placebo

SUMMARY:
The specific aim of this study is to examine the efficacy and safety of lisdexamfetamine compared with placebo in outpatients with binge eating disorder

ELIGIBILITY:
Inclusion Criteria:

* Patients will meet DSM-IV criteria for BED for at least the last 6 months

Exclusion Criteria:

* Women who are pregnant or lactating and women of childbearing potential who are not taking adequate contraceptive measures. If there is a possibility a female subject might be pregnant, a pregnancy test will be performed. (All women of childbearing potential will have a negative pregnancy test before entering the study.)
* Subjects who are displaying clinically significant suicidality or homicidality.
* A current or recent (within 6 months of the start of study medication) DSM-IV diagnosis of substance abuse or dependence

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
frequency of binge eating episode | 12 weeks
  frequency of binge eating episode

CONTACTS AND LOCATIONS:
Locations (1):
- Lindner Center of HOPE, Mason, Ohio, United States